CLINICAL TRIAL: NCT00131001
Title: Cost-Effectiveness Analysis of Imaging Strategies in Symptomatic Carotid Stenosis
Brief Title: CARMEDAS: Cost-Effectiveness Analysis of Imaging Strategies in Symptomatic Carotid Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 99.203
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2007-04

CONDITIONS: Carotid Stenosis
Keywords: Carotid artery stenosis; cost effectiveness; magnetic resonance angiography; computed tomography angiography; digital subtraction angiography
MeSH Terms: conditions — Carotid Stenosis

INTERVENTIONS:
Procedure: contrast-enhanced magnetic resonance angiography

SUMMARY:
PURPOSE: The purpose of this clinical trial is to study the cost-effectiveness ratios of diagnostic strategies for the imaging assessment of symptomatic carotid stenosis.

MATERIALS AND METHODS: The diagnostic accuracies of Doppler ultrasound (DUS), contrast-enhanced magnetic resonance angiography (CEMRA) and computed tomography angiography (CTA) were compared with digital subtraction angiography (DSA) in a multicenter study (CARMEDAS; 206 patients assessable) and in a meta-analysis (for CEMRA and CTA). The direct costs of each imaging method were calculated in 2 university medical centers. Eight hypothetical models were studied with DUS considered as the first-line imaging method and either CEMRA or CTA or DSA as the second or third line method. The effectiveness criterion was the number of potential avoided strokes for each strategy and for 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

Carotid artery stenosis > 50%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2001-04

PRIMARY OUTCOMES:
To study the cost-effectiveness ratios of diagnostic strategies for the imaging assessment of symptomatic carotid stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DOUEK, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France